CLINICAL TRIAL: NCT03124654
Title: Development and Validation of a Novel Educational Program for Patients Prescribed Non-vitamin K Anticoagulants (NOAC)
Brief Title: Development of a Questionnaire to Assess Patient Knowledge About Non-vitamin K Anticoagulants (NOAC)
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Other Study IDs: NOAC-Validation-study
Record Dates: First submitted 2017-04-07; First posted 2017-04-24 (Actual); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Atrial Fibrillation; Pulmonary Embolism; Deep Vein Thrombosis
MeSH Terms: conditions — Atrial Fibrillation; Pulmonary Embolism; Venous Thrombosis | interventions — Educational Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Education
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Patients will receive several questionnaires to fill in. Knowledge about NOACs will be assessed with a newly developped questionnaire and an educational program will be dispensed while analysing the answers (reactive educational program).

SUMMARY:
Pharmacists are in the best position to counsel and educate patients on anticoagulant agents such as NOACs. This should enable patients to play a more active role in their treatment and ultimately enhance adherence behaviour. However, educational elements should be targeted to knowledge. Thus, the investigators will develop and validate a questionnaire that can assess knowledge about NOACs

ELIGIBILITY:
Inclusion Criteria:

* Intake of a NOACs (Rivaroxaban, Edoxaban, Dabigatran, Apixaban)
* ≥18 years
* Able to give written Informed consent in German

Exclusion Criteria:

* NOACs for orthopaedic indication
* Dementia in medical history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a prescription for NOACs
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Validation of the new questionnaire assessed by questionnaire | measured once at visit 1 (baseline)
  Patients will rate on a 4-point likert scale feasibility, acceptability and comprehension of the new questionnaire immediately after the questionnaire had been filled in the first time.
Sensitivity of the new questionnaire | 7 days after visit 1, before and after the educational program
  Number of correct/incorrect answers measured at visit 2 before and after the educational program has been dispensed (7 days after visit 1)
Test retest validity of the new questionnaire | 7 days
  Number of correct/incorrect answers measured at visit 1 and 2 (0 respectively 7 days after visit 1)

SECONDARY OUTCOMES:
Patient's adherence assessed by questionnaire | 14 days
  change in adherence between visits 1 (baseline) and visit 3
Patient's satisfaction assessed by questionnaire | 14 days
  change in satisfaction between visits 1 (baseline) and visit 3
Patient's health literacy assessed by questionnaire | assessed once at visit 1 (baseline assessment)

OTHER OUTCOMES:
Number of patients having an anticoagulation identification card | assessed once at visit 1 (baseline assessment)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Hersberger, Prof., Study Chair — University of Basel; Isabelle Arnet, PD., Principal Investigator — Pharmaceutical Care Research Group, University of Base
Locations (1):
- University of Basel, Pharmaceutical Care Research Group, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No